CLINICAL TRIAL: NCT03541720
Title: 18F-Fluorodopamine PET Studies of Neuroblastoma and Pheochromocytoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLOPET; NCI-2018-01306 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2018-05-02; First posted 2018-05-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Neuroblastoma; Pheochromocytoma
MeSH Terms: conditions — Neuroblastoma; Pheochromocytoma | interventions — 6-fluorodopamine

STUDY DESIGN:
Intervention Model Description: 18F-DA scans will be performed within 4 weeks of standard imaging evaluations, such as CT (computed tomography) and I-123mIBG scanning.
  18F-DA will be injected into a vein in the arm or leg, or via central venous access line.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Injection of 18F-DA (Experimental): 18F-DA will be injected into a vein in the arm or leg, or via central venous access line.
  Interventions: Drug: 18F-DA

INTERVENTIONS:
Drug: 18F-DA — 18F-DA is an investigational PET radiotracer

SUMMARY:
PET (positron emission tomography) scans combined with a radioactive tracer will be used to identify and analyze tumors. Currently, the most common tracer used to analyze neuroblastoma tumors is called 123I-mIBG. However, the picture it provides is not always clear enough to see the very small areas of the disease.

18F-DA (18F-fluorodopamine) has been shown to be safe and more effective than 123I-mIBG in analyzing the tumor pheochromocytoma, which is closely related to neuroblastoma.

With this research study, the investigators plan to meet the following goals:

* Investigate to see if 18F-DA is safe to administer to pediatric patients with known or suspected neuroblastoma or pheochromocytoma
* Examine where in the body 18F-DA goes.
* Obtain information comparing 18F-DA to 123I-mIBG to see if 18F-DA could replace 123I-mIBG in the future.

About 20 people, with known or suspected neuroblastoma or pheochromocytoma, will take part in this Pilot study at St. Jude.

DETAILED DESCRIPTION:
Neuroblastoma is the most common extracranial malignant tumor of childhood. Nuclear imaging with 123I-mIBG is the standard test to follow and manage these patients. Because of the inherent imaging characteristics of I-123, there is suboptimal resolution within the images, causing them to appear somewhat blurry, which reduces our ability to find small areas of disease. A chemical that uses positron emission tomography should allow much better resolution of the images, which could improve patient care by allowing us to find small areas of disease that, if untreated, could result in tumor relapse. We have developed 18F-fluorodopamine (18F-DA) for PET imaging in our patients with neuroblastoma.

The primary objective is to explore the safety of 18F-DA in patients with known or suspected neuroblastoma or pheochromocytoma. The secondary objectives are to evaluate the biodistribution of 18F-DA in patients with neuroblastoma and compare the biodistribution of 18F-DA with the biodistribution of 123I-mIBG.

Patients receive an intravenous injection of a small (tracer) dose of 18F-DA. Approximately 1 hour later, patients undergo PET scanning of the entire body to evaluate the localization of the tracer.

ELIGIBILITY:
Inclusion Criteria:

Patients with known or suspected neuroblastoma or pheochromocytoma are eligible. 18F-DA PET/CT scanning will not be the initial imaging study in a newly diagnosed patient.

Patients with positive findings on prior imaging within the past 4 weeks are eligible.

Prior therapy is allowed.

Patients > 1 year of age, under the care of a SJCRH physician.

Patients of both genders, and all ethnic groups, under the care of a SJCRH physician.

Female participants of childbearing age must not be lactating due to theoretical potential harm to the infant from exposure to radiation.

Informed consent signed by participant, parent, or guardian according to the guidelines of the institutional review board.

Patients may undergo a repeat study one or more years following the initial FLOPET scan.

Exclusion Criteria:

Inability or unwillingness of patient, parent, or guardian to consent.

Pregnancy or lactation. Future plans for pregnancy do not exclude patient participation. Patients should not become pregnant within one month of completion of 18F-DA PET scan.

Use of medications known to interfere with 123I-mIBG uptake (principal considerations are phenylephrine and pseudoephedrine containing compounds which need to be discontinued for 48 hours, and labetalol which needs to be discontinued for 6 weeks).

Patients less than 3 years of age who require a total length of anesthesia time greater than 3 hours (for the FLOPET scan in conjunction with another clinical procedure requiring sedation) will be excluded from the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | up to 2 days following injection of the radiotracer 18F-DA.
  The adverse events will be recorded and monitored up to two days after the injection of radiotracer 18F-DA. The 95% CI for the adverse event rate will be calculated and reported. If one adverse event grade 2 or above, attributable to study drug, the study will be stopped until completion of IRB review and a decision about whether the study should be modified or closed.

SECONDARY OUTCOMES:
The frequency of localization of 18F-DA in different organs. | up to half year following injection of the radiotracer 18F-DA.
  The localization of 18F-DA throughout the whole body will be described descriptively in different organs such as salivary glands, heart, liver, kidneys, bladder, and bowel. The frequency of the localization of 18F-DA in those regions will be listed. Unexpected sites of uptake, such as bone or focally within soft tissue, are not normal and will be considered abnormal and documented descriptively as well.
max SUV from 18F-DA and 123I-mIBG PET | up to half year following injection of the radiotracer 18F-DA.
  Standardized uptake values of soft tissue and tumor (SUV) will be generated by drawing regions of interest on the images scaled to SUV. Descriptive statistics of SUV values, such as max SUV, from 18F-DA and 123I-mIBG PET will be provided.

OTHER OUTCOMES:
Mean and standard deviation of the difference of Curie scoring of 18F-DA and 123I-mIBG imaging | up to half year following injection of the radiotracer 18F-DA.
  The Curie scoring of 18F-DA and 123I-mIBG imaging will be scored for each participant. The difference of the Curie scoring between the two imaging will be calculated for each patient. Summary statistics of the difference such as mean and standard deviation would be calculated. One sample t test or signed rank test may be used to test whether the difference is equal to 0 depending on whether the distribution of the difference is normal or not.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Shulkin, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols